CLINICAL TRIAL: NCT02611635
Title: AF Patient Preferences Towards NOAC Versus VKA Treatment: a Patient Preference Study.
Brief Title: Atrial Fibrillation Patient Preference Study
Acronym: PRiSMA-AF
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18377
Record Dates: First submitted 2015-10-16; First posted 2015-11-23 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation
Keywords: non-valvular Atrial Fibrillation; Patient treatment preference; NOAC; VKA
MeSH Terms: conditions — Atrial Fibrillation | interventions — Vitamin B 6; Rivaroxaban

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VKA treatment of AF / Cohort 1: A sample of about 200 patients with non-valvular atrial fibrillation who are treated with VKAs for at least three months at date of study inclusion
  Interventions: Drug: VKA: Warfarin (Waran)
- NOAC treatment of AF / Cohort 2: A sample of about 200 patients with non-valvular atrial fibrillation who are treated with NOACs for at least three months at date of study inclusion
  Interventions: Drug: NOAC: Rivaroxaban (Xarelto, BAY59-7939); Drug: NOAC: Dabigatran etexilate; Drug: NOAC: Apixaban; Drug: NOAC: Edoxaban; Drug: NOAC: Lixiana

INTERVENTIONS:
Drug: VKA: Warfarin (Waran) — VKA have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: VKA treatment of AF / Cohort 1
Drug: NOAC: Rivaroxaban (Xarelto, BAY59-7939) — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: NOAC treatment of AF / Cohort 2
Drug: NOAC: Dabigatran etexilate — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: NOAC treatment of AF / Cohort 2
Drug: NOAC: Apixaban — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: NOAC treatment of AF / Cohort 2
Drug: NOAC: Edoxaban — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: NOAC treatment of AF / Cohort 2
Drug: NOAC: Lixiana — NOAC have been prescribed in the customary manner in accordance with the terms of the marketing authorization; decision to prescribe these agents has been made at least 3 months prior to study inclusion; assignment of a patient to a particular therapeutic strategy is only made retrospectively (treatment decision falls within current practice and the prescription of the medicines is separated from the decision to include the patient in the study)
  Groups: NOAC treatment of AF / Cohort 2

SUMMARY:
The main research question of this patient survey is to assess AF patients' preferences associated with different attributes which describe the different available anticoagulation treatment options (VKA or NOACs and, in case of NOACs, Apixaban, Dabigatran or Rivaroxaban).

VKA (Waran®) will be compared to Rivaroxaban.

DETAILED DESCRIPTION:
The objective of this study is to investigate the following research questions in a cross-sectional survey of Swedish AF patients being treated either with a VKA or with a NOAC:

* Which attributes of a medication to prevent stroke do AF patients view as important?
* Do AF patients have a preference regarding the attributes of the medication options VKA or NOAC and, in case of NOACs, with regards to rivaroxaban attributes?
* Are there subgroups of AF patients whose preference for one of the medication options appears above or below average?
* What is the quality of life of Swedish AF patients? Are there subgroups with differences in their quality of life (for example: subgroups of patients with different CHA2DS2-VASc scores)?
* Which burden do Swedish AF patients experience in association with their anticoagulation therapy? Are there differences in the burden of treatment (ACTS) between patients treated with VKA or with NOACs?

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for AF patients in both the NOAC and the VKA groups:

* Patients with a confirmed diagnosis of nonvalvular atrial fibrillation (persistent, paroxysmal, permanent),
* Age of at least 18 years at time of study inclusion,
* Generally willingness (informed consent) and ability to fill out a survey on satisfaction with treatment and quality of life, and to conduct a structured phone interview (approx. 20 - 30 min) in Swedish language.

Additional inclusion criterion for Group 1 (NOAC):

* Continuous anticoagulation with either Apixaban, or Dabigatran or Rivaroxaban for prevention of Stroke & systemic embolism for at least the previous 3 months.

Additional inclusion criterion for Group 2 (VKA):

* Continuous anticoagulation with a VKA for prevention of Stroke & systemic embolism for at least the previous 3 months.

Exclusion Criteria:

Exclusion criteria for both groups:

* Participation in another

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in primary care / internal medicine specialist practices or cardiology outpatient clinics in Sweden.
Sampling Method: Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
AF patients'preferences towards anticoagulation treatment with either VKAs or NOACs measured with a DCE (discrete choice experiment) design in a phone interview: Frequency of intake (once/twice daily) | up to 4 weeks after enrollment of patient
AF patients'preferences towards anticoagulation treatment with either VKAs or NOACs measured with a DCE (discrete choice experiment) design in a phone interview: Need of International normalized ratio (INR) monitoring/dose adjustment (yes/no) | up to 4 weeks after enrollment of patient
AF patients'preferences towards anticoagulation treatment with either VKAs or NOACs measured with a DCE (discrete choice experiment) design in a phone interview: Need of bridging (yes/no) | up to 4 weeks after enrollment of patient
AF patients'preferences towards anticoagulation treatment with either VKAs or NOACs measured with a DCE (discrete choice experiment) design in a phone interview: Interactions with food/drugs (yes/no) | up to 4 weeks after enrollment of patient
AF patients'preferences towards anticoagulation treatment with either VKAs or NOACs measured with a DCE (discrete choice experiment) design in a phone interview: Distance to treating physician (1km or 50km). | up to 4 weeks after enrollment of patient

SECONDARY OUTCOMES:
Patient-related burden of treatment with anticoagulants measured by the Benefit and Burden Scale of the Anti-clot Treatment Scale (ACTS) | Baseline
Patient's quality of life measured using the SF-12 (interview version) | up to 4 weeks after enrollment of patient
  Variables: Physical/psychological domain according to SF-12 questionnaire
Assessment of factors that may be associated with AF patients' preferences towards a specific anticoagulation treatment: Age | Baseline
Assessment of factors that may be associated with AF patients' preferences towards a specific anticoagulation treatment: Gender | Baseline
Assessment of factors that may be associated with AF patients' preferences towards a specific anticoagulation treatment: preferred Anticoagulation treatment (agent) | Baseline
Assessment of factors that may be associated with AF patients' preferences towards a specific anticoagulation treatment: HrQoL as defined by the SF-12 score | Baseline
Assessment of factors that may be associated with AF patients' preferences towards a specific anticoagulation treatment: AF symptoms as measured by the EHRA | Baseline
Assessment of factors that may be associated with AF patients' preferences towards a specific anticoagulation treatment: TTR (for VKA patients only) | Baseline
Assessment of factors that may be associated with AF patients' preferences towards a specific anticoagulation treatment: Lifestyle variables | Baseline
Assessment of factors that may be associated with AF patients' preferences towards a specific anticoagulation treatment: Previous switch of anticoagulation treatment | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Sweden